CLINICAL TRIAL: NCT06924086
Title: The Children's Adaptive Deep Brain Stimulation for Epilepsy Trial (CADET): a Pivotal, Randomized, Controlled, Double-blinded Multi-site Clinical Trial of Deep Brain Stimulation to Treat Children With Lennox-Gastaut Syndrome
Brief Title: The Children's Adaptive Deep Brain Stimulation for Epilepsy Trial
Acronym: CADET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); University of Oxford (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 141268
Record Dates: First submitted 2025-03-28; First posted 2025-04-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lennox Gastaut Syndrome (LGS)
Keywords: epilepsy; deep brain stimulation; Lennox-Gastaut Syndrome; pediatric; paediatric; children
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early stimulation (Active Comparator): Active stimulation
  Interventions: Device: Deep Brain Stimulation
- Delayed stimulation (Sham Comparator): Inactive stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Picostim DBS Device

SUMMARY:
The CADET Trial will investigate the effectiveness of deep brain stimulation (DBS) to reduce the frequency of seizures in children with Lennox-Gastaut syndrome (LGS). The CADET Trial will use a non-CE/UKCA marked device - the Picostim DBS system.

The SMART-DBS study is a sub-study of the CADET Trial. SMART-DBS will investigate the application of adaptive DBS for the treatment of children with LGS. Children will be recruited after they exit from either the prior 'CADET Pilot Study' or 'CADET Trial' - meaning that these children will already be receiving therapy with an already implanted Picostim device.

DETAILED DESCRIPTION:
All participants will complete a 4 week baseline assessment phase, then surgical implantation of the Picostim device and then a 4 week recovery phase. The participants will thereafter be randomised (1:1) and double-blinded to either an 'early stimulation' (DBS device switched on) or an 'delayed stimulation' (DBS device switched off) arm. Children allocated to receive early stimulation will complete 36 weeks of immediate active stimulation and children allocated to delayed stimulation will complete 12 weeks of inactive stimulation followed by 24 weeks of active stimulation.

The primary endpoint for all participants in the trial will be following 24 weeks of active stimulation. Secondary outcomes will be compared between the early and delayed stimulation arms following the first 12 weeks of the controlled phase.

The SMART-DBS study will recruit participants from the CADET Trial and the preceding CADET Pilot study. In both the CADET Trial and CADET Pilot studies, participants were fitted with the Picostim device and the device remains active. Participants who potentially meet the eligibility criteria will be provided with the PIS to consider participation in the adaptive DBS study.

ELIGIBILITY:
Children enrolled in this study must:

* Be 5-14 years of age at consent.
* Have a diagnosis of LGS, as determined by:

  * Slow (<3.0Hz) spike-and-wave pattern and/or fast wave pattern (tonic seizures) detected on EEG at least six-months prior to the enrolment into the baseline period
  * History of drop seizures (tonic, atonic, or tonic-clonic) that precedes at least six-months prior to the enrolment into the baseline period
* Have experienced at least 10 seizures in the four weeks prior to enrolment.
* Have tried and not responded to two or more antiseizure medications prior to enrolment.
* Be taking one or more anti-seizure medication(s) at a stable dose for at least the four weeks prior to enrolment.
* Have a carer who is willing for their child's maintenance anti-seizure medications and ketogenic diet (if relevant) to be unaltered for the trial duration.
* Have a carer who is willing and able to comply with all the requirements of the study, including the completion of the seizure diary and periodic device charging.

Children enrolled in this study must not:

* Have received prior deep brain stimulation insertion.
* Have an active ('on') vagus nerve stimulator (or active within the six months prior to the baseline period).
* Have had a change in their anti-seizure medication prescription or stopped their ketogenic diet within the last 4 weeks
* Have started or made changes to the prescription of a ketogenic diet within the last 12-weeks
* Have abnormal thalamic anatomy detected on imaging that would render DBS either unsafe or unfeasible.
* Have a bleeding disorder(s).
* Have a medical condition(s)/factor(s) that would increase their anaesthetic risk to an unacceptable level.
* Have a nickel allergy.
* Be pregnant.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency reduction | 24 weeks of active stimulation compared to baseline
  Seizure frequency reduction measured on carer-recorded seizure diaries

SECONDARY OUTCOMES:
Seizure frequency | 8-12 weeks following randomisation between the active and inactive stimulation arms
  Seizure frequency reduction measured on carer-recorded seizure diaries
Seizure frequency | 24 weeks of active stimulation compared to baseline
  Seizure frequency reduction measured on scalp EEG
Seizure frequency | 8-12 weeks following randomisation between the active and inactive stimulation arms
  Seizure frequency reduction measured on scalp EEG
Seizure severity | 24 weeks of active stimulation relative to baseline and comparison 12 weeks following randomisation between the active and inactive arms
  Seizure severity (according to the Hague Seizure Severity Scale). The HSSS scores range from 13 (least severe) and to 53 (most severe).
Quality of life (PedsQL) | After 24-weeks of active stimulation, and 12 weeks following randomisation between the active and inactive stimulation arms
  The PedsQL (Pediatric Quality of Life Inventory) questionnaire provides a quantitative score ranging from 0 (worst possible QoL) to 100 (best possible QoL) (https://www.pedsql.org/).
Quality of life (IPES) | After 24-weeks of active stimulation, and 12 weeks following randomisation between the active and inactive stimulation arms
  The Impact of Pediatric Epilepsy Scale (IPES) is a 12-item questionnaire that is answered by the carers of children with epilepsy that, as titled, aims to objectively measure the burden that epilepsy has on the child's life. The IPES scores range from 0 (lowest impact of epilepsy on the participant) to 33 (highest impact of epilepsy on the participant).

IPD SHARING:
Plan to Share IPD: Undecided